CLINICAL TRIAL: NCT04976608
Title: Relationship of Retinal and Visual Cortex Structure and Visual Acuity After Congenital Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: amblyopia-LZL
Record Dates: First submitted 2021-07-05; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Congenital Cataract
Keywords: amblyopia; MRI; SD-OCT; visual acuity; retinal structure; visual cortex structure
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: The BCVA of eyes is greater than 0.6
- Group 2: The BCVA of eyes is from 0.1 to 0.6
- Group 3: The BCVA of eyes is less than 0.6

SUMMARY:
To evaluate the influence of the visual acuity after congenital surgery on the retinal and visual cortex structure.

DETAILED DESCRIPTION:
According to the visual acuity after congenital cataract surgery, 30 patients are divided into 3 groups.SD-OCT and MRI were used to measure the parameters of the retina and the visual cortex, to compare the differences between different groups, and to analyze the relationship between the structure of the retina and the visual cortex and visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* age of 4-60 years
* Congenital cataract surgery is planned
* The operation was successful without any complications
* Can cooperate well with OCT and MRI examinations

Exclusion Criteria:

* Intraoperative and postoperative complications include glaucoma, retinal, corneal, or refractive medium diseases
* Behavioral, cognitive impairment
* Developmental delay

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with congenital cataract and were informed about their inclusion in the study and provided written consent.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Macular thickness | 2021.12.30
  Scan the 3.0mm diameter ETDRS ring area in the macular area with SD-OCT.
Subfoveal choroidal thickness | 2021.12.30
  Scan the Subfoveal choroid in enhanced scan mode with SD-OCT.
Retinal nerve fiber layer thickness | 2021.12.30
  Scan concentric circles with a length of 3.4mm and a diameter ranging from 2.5mm to 4.0mm in 12 directions centered on the optic disc with SD-OCT.
The volume of the lateral geniculate body | 2021.12.30
  Measure the volume of the lateral geniculate body by T1 phase scan of MRI
The volume of the brodmann 17,18,19 area | 2021.12.30
  Masure the volume of the brodmann 17,18,19 area by T1 phase scan of MRI
The FA of the white matter fiber bundle | 2021.12.30
  Measure the Fraction Anisotropy of the white matter fiber bundle related to visual signal transduction by DWI scan of MRI

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] Lu L, Li Q, Zhang L, Tang S, Yang X, Liu L, Sweeney JA, Gong Q, Huang X. Altered cortical morphology of visual cortex in adults with monocular amblyopia. J Magn Reson Imaging. 2019 Nov;50(5):1405-1412. doi: 10.1002/jmri.26708. Epub 2019 Mar 10. PMID 30854758
- [Background] Allen B, Schmitt MA, Kushner BJ, Rokers B. Retinothalamic White Matter Abnormalities in Amblyopia. Invest Ophthalmol Vis Sci. 2018 Feb 1;59(2):921-929. doi: 10.1167/iovs.17-22930. PMID 29450539
- [Background] Long E, Zhang X, Liu Z, Wu X, Tan X, Lin D, Cao Q, Chen J, Lin Z, Wang D, Li X, Li J, Wang J, Li W, Lin H, Chen W, Liu Y. Dynamic response to initial stage blindness in visual system development. Clin Sci (Lond). 2017 Jun 28;131(13):1515-1527. doi: 10.1042/CS20170234. Print 2017 Jul 1. PMID 28539328